CLINICAL TRIAL: NCT06149819
Title: Nurse Pathway for the Diagnosis of Non-traumatic Chest Pain in the Emergency Department: Preliminary Pilot Study (Chest Pain Nurse Track)
Brief Title: Chest Pain Nurse Track
Acronym: CHESTNUT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC22.0276; ID-RCB: 2023-A00058-37 (Other: National Agency for the Safety of Medicines and Health Products)
Record Dates: First submitted 2023-11-20; First posted 2023-11-29 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Chest Pain
Keywords: non traumatic chest pain; Nurse; management; track
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Intervention Model Description: This is a controlled, single centre, non-randomized, open-label interventional study evaluating the implementation of a nursing pathway management for chest pain. This study is an external comparison with a control group consisting of patients meeting the same eligibility criteria admitted to the Emergency Department over the same period and included prospectively with a 1:1 ratio. This design was chosen because of the difficulty of randomizing patients (few trained nurses) and the need to conduct a pivotal study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (paramedical) (Experimental): The patients will be cared for by one of the specially trained nurses based on a previously established allocation per day. A nurse will be able to take in charge several patients successively included on the same day, in accordance with the actual practice of organized intra-hospital sector and according to the standardized algorithm based on the recommendations.
  The DSMB will analyzed the compliance and safety of the management in this group at 20, 50 and 50% of enrollment and at the request of the sponsor if necessary.
  An adjudication committee will determine compliance with diagnostic management in the two groups.
  Interventions: Other: Diagnostic and safety of a nursing pathway for the management of non-traumatic chest pain
- Control (medical) (No Intervention): In this group the patients will received usual medical care over the same period in the emergency department and meeting eligibility criteria. Patients will be included prospectively after obtaining their consent, with a 1:1 ratio with sex and age correspondence +/- 5 years).
  An adjudication committee will determine compliance with diagnostic management in the two groups.

INTERVENTIONS:
Other: Diagnostic and safety of a nursing pathway for the management of non-traumatic chest pain — trained nurses will take in charge non-traumatic chest pain patient according to the standardized algorithm based on the recommendations .
  Arms: Intervention (paramedical)

SUMMARY:
Chest pain is a commonly encountered presentation in the emergency department (ED), with an incidence ranging from 5 to 12%. Chest pain has a wide range of aetiologies from the mildest to the most severe. In benign forms these pains can be musculoskeletal, psychogenic or even indeterminate (>60% depending on the place of recruitment). Coronary aetiology represents 12 to 25% of severe forms.

The management of chest pain in the emergency department is part of the daily life of nurses. According to the french 2020 Nurse Reception Organizer (IOA) guidelines, a nurse who has been trained for this role is required to "triage" (severity grade and orientation) patients presenting for this reason. The presence of specialized nurses in the management of chest pain allows faster initial management.

To date, no study has been conducted to assess the diagnostic and treatment performance of a nursing pathway for the management of patients presenting with acute chest pain regardless of the suspected diagnosis and not only acute coronary syndrome.

DETAILED DESCRIPTION:
The main objective of this interventional study is to evaluate the diagnostic safety of a nursing pathway for the management of patients presenting with chest pain in the emergency department compared with usual medical care.

This study is an external comparison with a control group consisting of patients meeting the eligibility criteria admitted to the Emergency Department over the same period and included prospectively with a 1:1 ratio.

The study will be conducted in three phases :

1. Training volunteer emergency department nurses (11) : the course will cover all aspects of management of non-traumatic chest pain (physiopathology, from diagnosis to treatment).

   For the selection of nurses, these criteria will need to be met : minimum of five years of practice in the profession with at least three years in emergency department ; the nurse must have had the training as a Nurse Reception Organizer and have received specific training in accordance with the study protocol.
2. Enrollment of 182 patients admitted to the emergency department for non-traumatic chest pain.

   The patient will be enrolled either in the experimental (paramedical) or control (medical) group. 91 patients will be included in each group.

   Experimental (Intervention) group or (paramedical cohort) :

   The patient is cared for by one of the specially trained nurses based on a previously established allocation per day. A nurse will be able to take in charge several patients successively included on the same day, in accordance with the actual practice of organized intra-hospital sector.

   The nurse will manage the patient according to the standardized algorithm based on the recommendations. An emergency physician will be systematically involved in the management process for interpretation of electrocardiogram (EKG) and chest x-ray, during a positive diagnosis, a sign of gravity and finally at any time as soon as the nurse considers it necessary. In addition each patient will be systematically examined and reassessed by a physician during paramedical management to validate the clinical, therapeutic and discharges conclusions.

   Control group (or medical cohort) :

   Cohort of patients receiving usual medical care over the same period in the emergency department and meeting eligibility criteria. Patients in this group will be included prospectively after obtaining their consent, with a 1:1 ratio with sex and age correspondence +/- 5 years).

   An independent adjudication committee comprising at least one emergency physician and one cardiologist will be responsible for analyzing the medical records of all patients (included in the two groups) in order to determine compliance with diagnostic management. It will meet before each Data and Safety Monitoring Board (DSMB) meeting (at 20, 50 and 80%) and at the end of the study.

   Data and Safety Monitoring Board (DSMB)composed of a methodologist, a cardiologist and an emergency physician. The DSMB will be responsible for analyzing the compliance and safety of management in the experimental group at 20, 50 and 80% of enrollment and at the request of the sponsor if necessary. This committee will also analyze the one month outcome of the patients included. It will decide whether to prosecute or stop the study.
3. Phone call follow-up of patient after one month to collect data :

   * Intercurrent serious events : death, re-admission, myocardial infarction, serious AE
   * Assessment of patient satisfaction
   * Any additional examinations and consultations carried out.

ELIGIBILITY:
Inclusion Criteria:

* Admission to emergency department (ED) for non-traumatic Chest Pain
* Affiliation to the French social security system
* Written informed consent must be obtained
* For women of childbearing age: effective contraception in place for at least 3 months. The absence of pregnancy should be confirmed by a negative urine test without delaying the start of the management including the realization of Electrocardiogram (EKG/ECG).

Exclusion Criteria:

* Suspected alcohol, drug or toxic intoxication
* Chest pain with associated neurological signs
* Patient with pacemaker or defibrillator
* Patient in vital distress requiring immediate medical intervention
* Patient admitted with a previously established aetiological diagnosis
* Unable to communicate or non-french speaking patients or those with impaired comprehension or consciousness
* Pregnant or breast-feeding patients
* Subject under administrative or judicial control, under protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who benefited from a diagnosis and overall management in accordance with medical recommendations in the paramedical group compared with usual medical care. | 30 days
  Rate of patients who benefited from a diagnosis and overall management in accordance with medical recommendations in the paramedical group compared with usual medical care after adjudication by an expert committee.

SECONDARY OUTCOMES:
Time in minutes between admission to emergency department and realization of Electrocardiogram (EKG/ECG | 15 minutes
  Time in minutes between admission to emergency department and realization of Electrocardiogram (EKG/ECG
Total duration in minutes of management in both cohorts between patient admission and effective patient discharge from emergency department. | 30 days
  Total duration in minutes of management in both cohorts between patient admission and effective patient discharge from emergency department .
All-cause care consumption in each cohort at one month | 30 days
  All-cause care consumption in each cohort at one month
Rate of Major Adverse Cardiovascular Events (MACE) at one month in each cohort | 30 days
  Rate of Major Adverse Cardiovascular Events (MACE) at one month in each cohort
Refusal rate of participation in the study in the paramedical cohort | 24 hours and 30 days
  Refusal rate of participation in the study in the paramedical cohort
Patient satisfaction assessed during discharge and at one month in both cohort | 24 hours and 30 days
  Patient satisfaction assessed during discharge and at one month by a numerical scale in both cohort numbered from 1 to 10 : (Not satisfied patient would no longer accept a nurse's care - Completely satisfied patient would accept to be cared for again by a nurse)
Assessment of quality of life during discharge and at one month in both cohort | 24 hours and 30 days
  Assessment of quality of life using EuroQol 5-dimension scale at discharge from emergency department and at one month in both cohort numbered from 0 to 100 : (the worst health you can imagine -the best health you can imagine)

CONTACTS AND LOCATIONS:
Overall Officials: Damien VIGLINO, Principal Investigator — Emergency Department of University Hospital Grenoble; Florian BARRET, Bachelor, Study Director — Emergency Department of University Hospital Grenoble; Karine FANJAS, Bachelor, Study Director — Emergency Department of University Hospital Grenoble
Locations (1):
- CHU Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: Yes
The international writing and publication rules (The Uniform Requirements for Manuscripts of the ICMJE, April 2010) will be followed. The minimum anonymized source data for performing the statistical analysis will be made public at the time of publication, with the article, or deposited in an appropriate public database. Other anonymized data may be available from the principal investigator upon reasonable request and with the consent of the sponsor.
  In accordance with the French law n ° 2002-303 of March 4, 2002, the subjects can be informed, at their request, of the overall results of the research. In this study, the investigators commit to individually communicating the overall results to each subject participating in the research by a short (popularized) summary and associated with a copy of the scientific article.
Supporting Information: Study Protocol, SAP
Time Frame: at the time of publication
Access Criteria: The international writing and publication rules (The Uniform Requirements for Manuscripts of the ICMJE, April 2010) will be followed. Moreover, In accordance with the French law n ° 2002-303 of March 4t, 2002